CLINICAL TRIAL: NCT04979754
Title: Long-term Renal Outcome After Cardiac Surgery : Impact of Previous Renal Transplantation
Brief Title: REnal TRansplant Outcomes After CARdiac Surgery (RETROCAR)
Acronym: RETROCAR
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Principal Investigator, Alexandre Ouattara, MD, PhD, University Hospital, Bordeaux
Other Study IDs: SAR Sud study one
Record Dates: First submitted 2021-07-05; First posted 2021-07-28 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass; Renal Transplant Recipient
Keywords: cardiac surgery; renal transplant recipient; renal function; acute kidney injury; major adverse kidney events
MeSH Terms: conditions — Acute Kidney Injury | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RENAL TRANSPLANT RECIPIENTS: All patients with previous renal transplantation undergoing cardiac surgery with cardiopulmonary bypass
  Interventions: Other: standard of care
- NON RENAL TRANSPLANT RECIPIENTS: All patients without previous renal transplantation undergoing cardiac surgery with cardiopulmonary bypass
  Interventions: Other: standard of care

INTERVENTIONS:
Other: standard of care — retrospective study : standard of care

SUMMARY:
In this retrospective study, the authors assess long term renal outcome in renal transplant recipients after cardiac surgery with cardiopulmonary bypass, and research factors associated with poor long term renal outcome.

DETAILED DESCRIPTION:
Post-operative mortality after cardiac surgery is increased in renal transplant recipients, compared with general population of cardiac surgery, or with kidney transplant recipients not undergoing cardiac surgery. If the survival of this specific population is now well studied, the long-term renal outcome is much less studied. Previous studies show a trend for increased risk of allograft dysfunction and need for permanent dialysis. This study proposes to compare long term renal outcome between renal transplant recipients and non-renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria for Renal Transplant Recipients group:

* Previous renal transplantation
* Who underwent cardiac surgery with CPB

Inclusion Criteria for Non Renal Transplant Récipients group:

* No previous renal transplantation
* Who underwent cardiac surgery with CPB
* Apparied with Renal Transplant récipients with the 5 following criteria : age, sex, previous diagnosis of diabete, type of cardiac surgery (isolated coronary artery bypass graft, valvular surgery, aorta surgery, combined surgery), best glomerular filtration rate with CKD-EPI formula at +/- 15 ml/min, in the 3 pre-operative months

Exclusion Criteria:

* Patients requiring mechanical circulatory support (Extracorporeal Membrane Oxygenation)
* Pre-operative permanent dialysis
* Aorta dissection extended to renal arteries
* Non-elective surgery for infective endocarditis
* Previous hepatic, pancreatic or cardiac transplantation
* Death in the 30 first days after cardiac surgery
* Patient not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive renal transplant récipients, apparied in a 1:2 ratio with non renal transplant récipients, undergoing cardiac surgery, and meeting the protocol criteria between january 2010 and december 2019, in university hospital of Bordeaux.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Long-term renal outcome | 12 months after surgery
  Proportion of patients meeting a composite criterion : death or permanent dialysis or doubling the baseline serum creatinine value

SECONDARY OUTCOMES:
Glomerular Filtration Rate (GFR) | 30 days after surgery
  Glomerular Filtration Rate (GFR) calculated with CKD-EPI formula
Glomerular Filtration Rate (GFR) | 12 months after surgery
  Glomerular Filtration Rate (GFR) calculated with CKD-EPI formula
Vital status | 12 months after surgery
  Mortality after surgery
Major Adverse Kidney Events | Up to 12 months after surgery
  Major Adverse Kidney Events defined by new receipt of Renal replacement therapy (RRT), or Acute Kidney Injury (AKI) episodes with persistent renal dysfunction and final serum creatinine value before hospital discharge ≥ 200 % of the baseline serum creatinine

CONTACTS AND LOCATIONS:
Locations (1):
- Bordeaux University Hospital, Pessac, France

IPD SHARING:
Plan to Share IPD: No